CLINICAL TRIAL: NCT03746665
Title: Maternal Immunization With MenAfriVac™
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Public Health England (Other Government); Department of State for Health and Social Welfare, The Gambia (Other Government); World Health Organization (Other); University of Cambridge (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SCC 1585
Record Dates: First submitted 2018-08-27; First posted 2018-11-20 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Meningitis; Meningococcal
Keywords: Men A; Maternal; Systems Immunology; Vaccination
MeSH Terms: conditions — Meningitis | interventions — MenAfriVac

STUDY DESIGN:
Intervention Model Description: 100 eligible mother-infant pairs randomized to the control group in the PROPEL trial (SCC1433, NCT02628886) who gave consent for their samples to be used for other ethically-approved research will be chosen at random and serve as controls for this study
Who Masked: Outcomes Assessor
Masking Description: Laboratory personnel assessing primary and secondary serological endpoints (Men A and Tetanus Toxoid) will be blinded to group allocation (i.e. MenAfriVac Group versus Control Group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- meningococcal serogroup A conjugate (Experimental): mothers will be vaccinated with meningococcal serogroup A conjugate vaccine between 28 - 34 weeks gestation
  Interventions: Biological: meningococcal serogroup A conjugate vaccine
- control (No Intervention): serological samples from 100 control mother-infant pairs already recruited as part of the PROPEL trial, (SCC1433), NCT02628886

INTERVENTIONS:
Biological: meningococcal serogroup A conjugate vaccine — Once final eligibility has been confirmed by a study clinician on the day, expectant mothers will be administered a single intramuscular dose of MenAfriVac™.
  Other Names: MenAfriVac™.
  Arms: meningococcal serogroup A conjugate

SUMMARY:
The World Health Organization (WHO) recommends that infants receive a single dose of the meningococcal serogroup A-tetanus toxoid conjugate vaccine, MenAfriVac, when they reach at least 9 months of age. However, this leaves a window of susceptibility in early life when the incidence of invasive serogroup A disease, and the case fatality rate for the condition is at its highest. This study will investigate the potential role of administering the vaccine to expectant mothers at the start of the third trimester of pregnancy in order to protect their subsequent borne infants. Antibody transfer to the newborn and subsequent antibody decay will be measured. The level of protection against neonatal tetanus provided by the tetanus toxoid component of the vaccine, when compared to the routine dose of tetanus administered in pregnancy will also be assessed.

As a separate exploratory study, the follow-up of the cohort planned will also be used to investigate the effects that the development of the gastrointestinal microbiome, and any perturbations in the microbiome caused by antibiotic use, have on immune development and vaccine immunogenicity over the first 10 months of life.

DETAILED DESCRIPTION:
MenAfriVac is a Neisseria meningitidis serogroup A Men A polysaccharide-tetanus toxoid conjugate vaccine which was developed within the space of just nine years through the Meningitis Vaccine Project. Although the effectiveness of the vaccine is well established, the optimum strategy for maintaining protection following the mass vaccination campaigns has yet to be determined. However, in mathematical models, even considering a coverage rate of as low as 60 percent, the routine administration of MenAfriVac nine-months results in a lower annual disease incidence than regular campaigns targeting one to four year old children. Thus, the introduction of a single dose of MenAfriVac® at nine to 18 months in meningitis belt has subsequently been recommended by the WHO.

An important limitation of such a regimen is that infants are left without direct protection against Men A infection up to the age of at least nine months. While not classically considered to be a disease of early infancy, the incidence of invasive Men A infection is as high or higher in this age group as compared to the incidence in older children and the case fatality rate is also at its peak under the age of one. Recent mass vaccination campaigns rapidly achieved exceptionally high levels of coverage across the entire one to 29 year old adult population and have resulted in herd protection and reduced level of invasive disease in those under one year of age. However, such levels of herd protection cannot be assumed following routine scheduling at nine months of age and thus alternative strategies both to protect the infant up to nine months of age and also to boost herd protection in the population warrant exploration.

Maternal immunization represents a potentially attractive option with both regards. The safety of the vaccine when administered in pregnancy has been assessed through comparing the rate of safety events in 1730 expectant mothers immunized during campaigns in the Navrongo region of Ghana, and their subsequent born infants with the rates in the women who did not receive the vaccine during the same campaign (n=919) and those vaccinated the previous year (n=3551). No evidence of any safety concerns were reported. These data support current WHO technical guidance which considers it safe to include pregnant and lactating women within mass vaccination campaigns. Although the safety profile is reassuring, there are currently no data on the immunogenicity of MenAfriVac in pregnancy or on the transplacental transfer of Men A specific antibodies to subsequent borne infants. In addition, the comparability of the tetanus toxoid specific seroprotection provided to the newborn through the tetanus toxoid carrier protein and through the standard tetanus toxoid antenatal booster needs to be established.

Within the Protecting from Pneumococcus in Early Life (PROPEL) trial (NCT02628886) trial a group of 200 expectant mothers were randomized into the control group and received tetanus toxoid (and a 0.9% sodium chloride injection to maintain blinding) at 28 to 34 weeks gestation. This group will serve as a control group for the MenAfriVac vaccinated mothers who will be recruited here using an otherwise identical protocol. Those mothers confirmed to be eligible (n = 100) will receive a dose of MenAfriVac at 28 to 34 weeks of gestation and will subsequently followed up using the same approach as undertaken in the PROPEL trial. Their subsequent born infants will also be followed until nine months of age in the same way. Maternal and cord blood samples will be collected at delivery with peripheral infant samples being obtained at delivery, 8 and 20 weeks and at 9 months plus 9 months 4 weeks. The meningococcal serogroup A and tetanus toxoid specific seroprotection in the infants of mothers vaccinated with MenAfriVac will be compared to the seroprotection in those mothers in the control group for the main randomized trial who will only have received tetanus toxoid in pregnancy. All safety procedures will be undertaken in the same way for comparability.

Most mothers in the study will have been immunized in the national MenAfriVac campaign in the Gambia in Nov/Dec 2013, so the controls will not be naïve, and the MenAfriVac arm will be receiving a second dose of the vaccine. This reflects the likely situation were maternal immunization to be recommended in the future. Information on prior immunization history will be collected and assessed within the statistical analysis.

Exploratory nested study:

The study provides an opportunity to monitor the development of the intestinal microbiome from birth to 10 months of age and to assess the effects that any antibiotics, administered in early life for clinical indication, have on this development. Furthermore, to study the downstream effects of distinct microbial profiles on baseline and post-vaccination transcriptomic and metabolomic profiles and immune cell phenotypes, and on the serological responses to vaccination.

The gastrointestinal microbiome is at its most dynamic in early life from the point of first colonization at birth. It is also the period during which parenteral empirical antibiotics are most likely to be administered given the difficulty in excluding invasive bacterial diseases at this age. Thus, early infancy provides the best possible opportunity to study the effects of the microbiome, including of any disruption in the microbiome driven by antibiotic therapy, on baseline (unstimulated) and post-vaccination transcriptomic and metabolomic profiles, immune cell phenotypes and serological response to vaccination.

This component of the study is observational and exploratory. All 100 infants will be administered the routine vaccines in the national schedule due at the time points they are routinely given. Associations between the development of the microbiome with transcriptional and metabolomics signatures, cellular and serological responses to vaccination will be made within group.

ELIGIBILITY:
Inclusion Criteria:

* Signed/thumb-printed informed consent for trial participation obtained*
* Pregnant woman aged between 18 and 40 years of age inclusive* (note that those over 33 years of age would not be expected to have been vaccinated in the national MenAfriVac™ campaign targeting 1 to 29 years olds in Nov/Dec 2013)7
* Singleton pregnancy*
* From 28 to 34 weeks gestation as determined by ultrasound scan
* Resident within easy reach of the clinical trial site (no fixed boundaries will be set, and such judgements will be made on a case by case basis by members of the field team in discussion with the potential participant, taking into account knowledge of the local transport links and geography) *
* Intention to deliver at the health centre related to the clinical trial site (i.e. Faji Kunda health centres) *
* Willingness and capacity to comply with all the study procedures, including those relating to the newborn infant, in the opinion of the principal investigator or delegee

Exclusion Criteria:

* History of pre-eclampsia or eclampsia*
* History of gestational diabetes*
* Rhesus negative multigravida who did not receive anti-D in previous pregnancies
* Five or more previous pregnancies (grand-multigravida)
* Previous late stillbirth (defined as loss of pregnancy at any time after 28 weeks gestation) *
* Previous premature delivery (defined as delivery before 37 weeks gestation) *

  • Previous neonatal death (defined as death of an infant within the first 28 days of life) *
* Previous Caesarean section*
* Previous delivery of an infant with major congenital anomalies (see Table 7 for definition) *
* Previous delivery of an infant with a known or suspected genetic9 or chromosomal abnormality*
* History of other significant pregnancy related complications judged likely to affect the safety of the mother or infant or to significantly compromise the endpoint data collected*
* History of other significant neonatal complications judged likely to affect the safety of the mother or infant or to significantly compromise the endpoint data collected*
* Significant complications in current pregnancy
* Significant alcohol consumption during current pregnancy
* Significant maternal chronic illness including but not limited to hypertension requiring treatment, heart disease, lung disease, neurological disorders including a history of epilepsy or recurrent afebrile seizures, kidney disease, liver disease, anaemia and other haematological disorders, endocrine disorders including known diabetes mellitus, autoimmunity
* Severe anaemia (<7.0g/dL) [35] *
* Known Human Immunodeficiency Virus (HIV) or hepatitis B (HBV virus positive or found to be HIV or HBV positive during screening*
* Positive result for syphilis infection on laboratory testing*
* Receipt of any vaccine during the current pregnancy or plans to receive any non-study vaccines during the current pregnancy (tetanus toxoid vaccination is not an exclusion and vaccines given during national campaigns if applicable will not generally be exclusions)
* Any other condition judged to significantly increase the risks to either the mother or the infant within the current pregnancy (including relevant history from previous pregnancies)
* History of anaphylactic or severe allergic reactions to previous vaccines or history of anaphylactic or severe allergic reactions in previous offspring (if applicable) *
* Receipt of any blood product including human immunoglobulins at any stage during the current pregnancy or plan to receive any blood products during the period of trial participation (receipt or blood products in an emergency or for obstetric reasons will not represent a protocol deviation given such situations are unplanned)
* Receipt of immunosuppressive or immuno-modulatory medication at any stage during the current pregnancy or plan to receive any such medication during the period or trial participation
* Clinically suspected or confirmed congenital or acquired clotting or bleeding disorders or the current receipt of medications known to alter clotting or bleeding*
* Current malaria infection (on the day of vaccination)
* Any clinically significant signs or symptoms of acute illness, significant abnormalities in vital signs, an axillary temperature of > 37.5°C or any recorded fever (> 37.5°C) in the preceding 24 hours.
* 2 or more symptoms (nausea/vomiting, diarrhoea, headaches, fatigue and myalgia) rated as grade 2 and clinically significant on the maternal systemic reactogenicity scale (Table 5) present at baseline on the day of vaccination

In cases on uncertainly, the clinical significance of any particular complaint will be judged by the PI, in discussion with other members of the clinical trial team. The safety of the expectant mother and unborn infant will always represent the key criteria with this regard. The basis of such decisions will be documented in the participant notes maintained by the clinical trial team.

In the case of an acute illness, including malaria, documented fever or abnormalities in vital signs, and also when 2 or more grade 2 systemic reactogenicity symptoms are present, the potential participant will not be deemed to be a screen failure and thus will not be permanently excluded from participation (unless the assessing clinician has reason be believe the problem will persist). Under these circumstances the expectant mother will be termed a temporary exclusion and will be re-screened at an appropriate interval for eligibility (a minimum of 24 hours in the case of a recorded fever and otherwise according to the clinical judgement of the clinician). If 34 weeks gestation passes during this period of observation, if any other inclusion criteria is no longer met (e.g. the potential participant reaches her 41st birthday) or if another exclusion criteria is met (e.g. the potential subject develops pre-eclampsia), the participant will be deemed to be a screen failure. Repeat serological testing for HIV, Hepatitis B and syphilis is not required at re-screening unless the PI has specific reason to believe that a potential participant's status may have changed in the interval since the original test. A repeat haemoglobin level is not required although may be undertaken if judged to be warranted on the basis of clinical assessment.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 200 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Meningococcal serogroup A (Men A) serum bactericidal activity (SBA) Geometric Mean Titre (GMT) | Infants at birth
Men A SBA GMT | Infants at 8 weeks of age
Men A SBA GMT | Infants at 20 weeks of age
Men A SBA GMT | Infants at 9 months of age
Percentage tetanus toxoid seroprotection | Infants at birth
Number of serious adverse events (SAE) in expectant mothers | Between 28 to 34 weeks gestation until 8 weeks from the end of pregnancy
Number of SAE in infants | From birth until 9 months of age
Injection site pain in mothers | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Injection site pain in infants | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Injection site tenderness in mothers | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Injection site tenderness in infants | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Injection site erythema in mothers | Day 1 to day 7 following vaccine administration
  Diameter of erythema in millimetres
Injection site erythema in infants | Day 1 to day 7 following vaccine administration
  Diameter of erythema in millimetres
Injection site induration in mothers | Day 1 to day 7 following vaccine administration
  Diameter of induration in millimetres
Injection site induration in infants | Day 1 to day 7 following vaccine administration
  Diameter of induration in millimetres
Axillary temperature in mothers | Day 1 to day 7 following vaccine administration
  Degrees Centigrade
Axillary temperature in infants | Day 1 to day 7 following vaccine administration
  Degrees Centigrade
Vomiting in mothers | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Vomiting in infants | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Diarrhoea in mothers | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Diarrhoea in infants | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Headaches in mothers | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Reduced feeding in infants | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Fatigue in mothers | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Drowsiness in infants | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Myalgia in mothers | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Irritability in infants | Day 1 to day 7 following vaccine administration
  Grade 0 to 5 severity
Pregnancy outcome | At delivery (approximately 40 weeks gestation)
  Late pregnancy loss, early stillbirth, late stillbirth, livebirth

SECONDARY OUTCOMES:
Men A immunoglobulin G (IgG) Geometric Mean Concentrations (GMC) | Infants at birth
  International units/millilitre
Men A GMC | Infants at 8 weeks of age
  International units/millilitre
Men A GMC | Infants at 20 weeks of age
  International units/millilitre
Men A GMC | Infants at 9 months of age
  International units/millilitre
Men A SBA GMT | Mothers at 28 to 34 weeks gestation
Men A SBA GMT | At delivery (approximately 40 weeks gestation)
Tetanus Toxoid IgG GMC | Infants at birth
  International units/millilitre
Tetanus Toxoid IgG GMC | Infants at 8 weeks
  International units/millilitre
Tetanus Toxoid IgG GMC | Infants at 20 weeks
  International units/millilitre
Tetanus Toxoid IgG GMC | Infants at 9 months
  International units/millilitre
Tetanus Toxoid IgG GMC | At delivery (approximately 40 weeks gestation)
  International units/millilitre
Men A immunoglobulin A levels in breast milk | 8 weeks from the end of pregnancy
  Units/millilitre
Men A immunoglobulin G levels in breast milk | 8 weeks from the end of pregnancy
  Unit/millilitre
Number of adverse events (AE) in expectant mothers | 28 to 34 weeks gestation until 8 weeks from the end of pregnancy
Number of AE in infants | From birth until 9 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Ed Clarke, MBChB, Principal Investigator — MRC @ LSHTM
Locations (1):
- Medical Research Council Unit (MRC), The Gambia, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: No